CLINICAL TRIAL: NCT04899895
Title: Rheumatology Biorepository
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: BIO-100
Record Dates: First submitted 2021-05-03; First posted 2021-05-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Biorepository is a prospective observational cohort study for patients under the care of a licensed physician or qualified physician extender. Target minimum enrollment is approximately 3,000 patients within the first 5 years of the study with no defined upper limit of enrollment. Sites from Corrona's current North America network will be asked to participate.

Participating sites and subjects will not receive results from any laboratory testing conducted on the Samples. Personal identifying information will not be collected along with the Samples.

Subjects will provide informed consent to contribute Samples to include blood (serum, plasma, whole blood) to the Biorepository. In the future, Subjects may be asked to contribute other samples (i.e. saliva, urine, stool) and an additional informed consent will be obtained. Subjects will retain the right to withdraw their consent for use of their Samples at any time. In such case, Corrona will destroy any unused/remaining Samples in its possession.

DETAILED DESCRIPTION:
The purpose of the study is to develop a biorepository of biological samples ("Samples") from eligible patients enrolled in the Corrona Rheumatology Registries (each, a "Registry", together the "Registries"), including but not limited to registries related to rheumatoid arthritis (RA), psoriatic arthritis and spondyloarthritis (PsA/SpA), osteoarthritis, and lupus (the "Biorepository"). Collected Samples will be biobanked for immediate or future analysis.

The Biorepository will be used for various purposes, including to support identification and validation of biomarkers predictive of drug toxicities, safety outcomes (e.g. infections, malignancies, autoimmunity, venous thromboembolism), or response to specific therapies used for the diseases studied in the Registries. Other objectives may include research on biomarkers that describe disease activity or phenotypic disease subsets, and research to understand mechanism of disease or comorbidities.

A wide array of testing methods may be used, such as DNA and RNA sequencing, targeted analysis to analyze protein, lipid, metabolite, small molecule or biologic assays, and/or other studies. Analysis of Samples may include testing for existing and commercially available laboratory measures or experimental analysis. Samples will be selected for testing depending on factors such as: the disease under study, qualifying treatment and/or cohort, patient characteristics, risk factors or disease activity indicators, and research questions.

The Biorepository study will seek to support research in various rheumatologic disease states through Sample analyses.

ELIGIBILITY:
A patient must satisfy all of the following criteria to be eligible for enrollment in the Biorepository study .1)Patient is currently participating in a Registry or is eligible to participate and enrolls in a Registry prior to enrollment in the Biorepository study.

2)Patient is starting an Eligible Medication*with no prior exposure to the specific medication being prescribed.

3)Patient is able to complete Sample collection within fourteen (14) days prior to receiving thefirst dose of the Eligible Medication.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The following eligibility criteria are designed to select patients for whom study assessments are deemed appropriate. Patients must have attained at least the locally recognized age of consent and provide written or electronic informed consent to participate
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
1. Biospecimen (blood) Collection | every 6 months for 10 years
  Establish a collection of blood samples from patients with Rheumatoid Arthritis
2. Laboratory testing | every 6 months for 10 years
  Testing for Biomarkers that describe disease activity or phenotypic disease subsets, risk prediction for certain types of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Corrona, LLC, Waltham, Massachusetts, United States